CLINICAL TRIAL: NCT03382587
Title: An Observational Study to Assess the Use of Intravitreal Aflibercept Injections in a Routine "Treat and Extend" Regimen in Treatment-naïve Patients Diagnosed With Wet Age-related Macular Degeneration
Brief Title: Observational Study to Assess Intravitreal Aflibercept Injections Used in a "Treat and Extend" Regimen in Treatment-naïve Wet Age-related Macular Degeneration Patients
Acronym: ASTERIA
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 18574
Record Dates: First submitted 2017-12-11; First posted 2017-12-26 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Wet Age-related Macular Degeneration
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aflibercept: Treatment-naive wet age-related macular degeneration patients under routine intravitreal aflibercept treatment in a treat-and-extend scheme
  Interventions: Drug: Aflibercept (Eylea, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, BAY86-5321) — Intravitreal aflibercept injections used in a routine "treat and extend" regimen, under which the intervals between the injections are extended if disease stability is maintained and no signs of worsening disease are observed on the injection day

SUMMARY:
The purpose of this observational study lies in the analysis of a treat-and-extend injection scheme with intravitreal aflibercept (i.e. injection into the eye), as applied in routine practice in previously untreated patients diagnosed with wet age-related macular degeneration.

DETAILED DESCRIPTION:
Data will be collected from the medical files retro- and prospectively. If patients are still under treatment at study initiation and have not yet completed 24 months of treatment with intravitreal aflibercept in a treat-and-extend regimen, data of the remaining observation period will be collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of wet age-related macular degeneration.
* No prior therapy for wet age-related macular degeneration.
* Patients for whom the decision to initiate treatment with IVT-AFL in a T&E regimen was made as per routine clinical practice.
* Patient age >55 years of age

Exclusion Criteria:

* Participation in an investigational program with therapeutical interventions outside of clinical routine practice.
* Patients with eye diseases e.g. advanced glaucoma or visually significant cataracts, likely to require surgery during the observation period in the study eye.
* Concomitant ocular or systemic administration of drugs up to 3 months before commencement of IVT-AFL treatment that could interfere with or potentiate the mechanism of action of aflibercept, including anti-VEGF agents. This includes patients receiving a different anti-VEGF agent for the fellow eye

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Treatment-naive wet age-related macular degeneration patients under routine intravitreal aflibercept treatment in a treat-and-extend scheme
Sampling Method: Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-27 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in best-corrected visual acuity in Early Treatment Diabetic Retinopathy Study letters (ETDRS letters) | Baseline and at 12 months
  mean change in ETDRS letters

SECONDARY OUTCOMES:
Mean change from baseline in best-corrected visual acuity (in Early Treatment Diabetic Retinopathy Study (ETDRS) letters) | Baseline and at 24 months
  mean change in ETDRS letters
Mean change in best-corrected visual acuity in relation to the number of injections administered | Baseline and at 12 months; Baseline and at 24 months
  Numbers of injections will be predefined as categories and analyzed in relation to the BCVA changes
Mean interval between injections | At 12 and 24 months
  mean interval displayed in weeks or days
Reasons for the interval length | At 12 and 24 months
  morphology and / or BCVA /other
Frequency of disease reactivation | Baseline and at 12 months; Baseline and at 24 months
  Disease activity such as hemorrhage, PED, subretinal fluid, cystoid intraretinal fluid, RPE rip assessed at the investigator's discretion as: none / new or increasing / decreasing / stable
Proportion of eyes gaining or losing ≥ 15 Early Treatment Diabetic Retinopathy Study letters compared to baseline | Baseline and at 12 months; Baseline and at 24 months
  Proportion evaluated as percentage (%) of eyes
Mean changes from baseline in central retinal thickness (CRT) | Baseline and at 3 months; Baseline and at 12 months; Baseline and 24 months
  micro meter (µm)
Changes from baseline in retinal fluid | Baseline and at 12 months; Baseline and at 24 months
  intraretinal or subretinal fluid or pigment epithelial detachment (PED)
Reasons for termination of therapy (including subsequent therapy at time of discontinuation) | At 12 and 24 months
  Categorized into typical reasons for discontinuation such as e.g. death, lost to Follow-up, withdrawal of informed consent, change of treatment regimen, discontinuation of IVT-AFL treatment, interfering surgery or treatment, adverse event, other
Severity of disease reactivation | Baseline and at 12 months; Baseline and at 24 months
  Severity of disease reactivation assessed at the investigator's discretion as: no new disease activity / mild / severe

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Multiple Locations, Switzerland

IPD SHARING:
Plan to Share IPD: No